CLINICAL TRIAL: NCT05275387
Title: the Effect of AQP-1 Polymorphism on Fluid Status of Hemodialysis Patients
Brief Title: AQP-1 Polymorphism on Fluid Status in Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Zanzhe Yu, Prinical Inverstigator, RenJi Hospital
Other Study IDs: KY2021-149-B
Record Dates: First submitted 2022-01-17; First posted 2022-03-11 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: End Stage Renal Disease on Dialysis
Keywords: AQP1; fluid status
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — total blood sample stored in local biospecimen facility
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational study, no intervention — observational study, no intervention

SUMMARY:
It is a cross sectional observational study. It is to investigate whether AQP-1 polymorphism has any impact on fluid status in hemodialysis patients. The long term stable HD patients in the current center will be enrolled to the study after informed consent. Blood samples will be collected for gene-typing. Fluid status including blood pressure, weekly UF and intra-dialysis body weight change will be collected through their clinical records.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70
* ESRD
* maintained HD
* no target weight change during the last week of entering the study and achieve target weight at the end of HD section
* informed consented

Exclusion Criteria:

* expected survival time less than 3 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ESRD patients on maintained hemodialysis.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
The total ultrafiltration volume in mls from hemodialysis for the whole week of the recruitment | up to 12 weeks
  The ultrafiltration volume of each HD section of the enrollment week will be recorded. The total ultrafiltration volume of the week is the primary outcome measure. (In most cases, HD patients have three HD sections per week.)

SECONDARY OUTCOMES:
The total weight gain in kgs of each HD section of the enrollment | up to 12 weeks
  The body weight gain of each HD section of the enrollment week will be recorded. The total body weight gain of the week is the secondary outcome measure. (In most cases, HD patients have three HD sections per week.)

CONTACTS AND LOCATIONS:
Overall Officials: Zanzhe Yu, PhD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided